CLINICAL TRIAL: NCT02777658
Title: PANORAMA - Real World Molecular Testing, Treatment Patterns, and Clinical Outcomes in Patients With EGFR Mutation-Positive Locally Advanced or Advanced NSCLC
Brief Title: PANORAMA - Real World Molecular Testing, Treatment Patterns, and Clinical Outcomes EGFR Mutation-Positive NSCLC
Acronym: PANORAMA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: iOMEDICO AG, Freiburg, Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: D5160R00005
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Epidermal Growth Factor Receptor (EGFR), non-small cell lung cancer (NSCLC), EGFR T790M, EGFR Mutation-Positive Locally Advanced or Advanced NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary Study Cohort: Patients with prior confirmed EGFR mutation-positive locally advanced or advanced NSCLC (Non-Small Cell Lung Cancer) who have progressed on or after EGFR-TKI (Epidermal Growth Factor Receptor - Tyrosine Kinase Inhibitor) therapy
- Secondary Study Cohort: Patients diagnosed with de-novo (wild-type) EGFR T790M mutation-positive (alone or in combination with other mutations) locally advanced or advanced NSCLC

SUMMARY:
The objectives of this study are to assess molecular testing, treatment patterns, and associated outcomes among patients with EGFR (Epidermal Growth Factor Receptor) mutation-positive locally advanced or advanced NSCLC (Non-Small Cell Lung Cancer) who have progressed on or after EGFR-TKI (EGFR-Tyrosine Kinase Inhibitor) therapy post availability of a third-generation TKI (primary study cohort). Additionally, molecular testing and treatment patterns will be assessed among a secondary cohort of patients which will include patients diagnosed with de-novo EGFR T790M mutation-positive locally advanced or advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria - Primary Study Cohort

* Provision of written informed consent (patient consent should be within 6 weeks of disease progression, defined elsewhere as the Index Date)
* Adult male or female subjects (according to age of majority/adulthood as defined by local regulations)
* Patients with prior confirmed EGFR mutation-positive (all mutations) locally advanced or advanced NSCLC - Patients who developed resistance to an EGFR-TKI due to any other phenotypic/histologic transformations (e.g., small-cell lung cancer, EMT) or other mutations (e.g., HER2, MET amplifications) at the index-date will be eligible for participation in this study as long as they have prior confirmed diagnosis of EGFR mutation-positive (all mutations) locally advanced or advanced NSCLC
* Patients who have progressed on or after EGFR-TKI therapy (i.e., gefitinib, erlotinib or afatinib) within the patient selection period

Inclusion Criteria - Secondary Study Cohort

* Provision of written informed consent (patient consent should be within 6 weeks of NSCLC diagnosis, defined elsewhere as the Index Date)
* Adult male or female subjects (according to age of majority/adulthood as defined by local regulations)
* Patients diagnosed with de-novo EGFR T790M mutation-positive locally advanced or advanced NSCLC during the patient selection period. The de-novo T790M mutation can be alone or in combination with other mutations (e.g., L858R and T790M).

Exclusion Criteria - Primary and Secondary Study Cohorts

• Enrollment in studies that prohibit any participation in this non-interventional study. These patients will be censored.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 800 patients across both cohorts - 700 patients primary cohort and 100 patients secondary cohort. Patients will be recruited from approximately 100 participating sites in Germany (70 hospitals and 30 outpatient practices).
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
To evaluate molecular testing patterns among patients with EGFR mutation-positive locally advanced or advanced NSCLC | Date of enrollment in the study until end of follow-up or death if this occurs before, assessed approximately up to 36 months
  Molecular testing patterns including:
  Molecular testing rate defined as the number of patients identified as having received molecular testing divided by the number of patients in the primary study cohort (applicable to patients in the primary study cohort);
  Change in testing rates over time - testing rate over time will be described;
  Molecular testing details including sample type, method of biopsy, testing turnaround time, test type, reason for testing, testing laboratory type, reason for not performing a test;
  Molecular testing results including mutation status and type, test outcome, histologic/phenotypic transformation;
To assess treatment patterns and associated clinical outcomes among patients with EGFR mutation-positive locally advanced or advanced NSCLC | Date of enrollment in the study until end of follow-up or death if this occurs before, assessed approximately up to 36 months
  Treatment patterns and associated clinical outcomes including:
  Overall survival measured from: date of initial diagnosis to date of death from any cause (for primary and secondary cohorts), date of progression to date of death from any cause (for primary cohort only);
  Time to initiation of new therapy defined as the time from start date of current therapy to start date of subsequent therapy;
  Treatment(s) received post diagnosis and post progression including chemotherapy, radiation, surgery, targeted therapy, immunotherapy; Treatment sequence patterns, line(s) of therapy, treatment regimen(s), treatment duration, number of cycles;

SECONDARY OUTCOMES:
To assess health care utilization patterns | Date of enrollment in the study until end of follow-up or death if this occurs before, assessed approximately up to 36 months
  Health care utilization patterns will be presented by the following care settings: hospitalization and length of stay, emergency room and physician office visits
To assess treatment related complications | Date of enrollment in the study until end of follow-up or death if this occurs before, assessed approximately up to 36 months
  Assessment of treatment related complications observed with chemotherapy and targeted therapies among patients with NSCLC.
To assess biopsy related complications | Date of enrollment in the study until end of follow-up or death if this occurs before, assessed approximately up to 36 months
  Assessment of biopsy related complications for each documented biopsy procedure
To document rate of central nervous system (CNS) metastases | Date of enrollment in the study until end of follow-up or death if this occurs before, assessed approximately up to 36 months
Assessment of health-related quality of life (HRQoL) | Date of first visit to last visit. HRQoL are collected every 6 months (plus or minus 1.5 months) up to 36 months
  Health related quality of life (HRQoL): Assessment of general cancer-associated and specific lung cancer associated parameters by use of standardized HRQoL questionnaires:
  * European Organization For Research And Treatment Of Cancer Quality Of Life Questionnaire - Core 30 (EORTC QLQ-C30)
  * European Organisation For Research And Treatment Of Cancer Quality Of Life Questionnaire - Lung Cancer 13 (EORTC QLQ-LC13) (adminstered to patients included in primary study cohort)

CONTACTS AND LOCATIONS:
Locations (73):
- Germany (73):
  - Research Site, Aschaffenburg
  - Research Site, Augsburg
  - Research Site, Bad Kreuznach
  - Research Site, Ballenstedt
  - Research Site, Bautzen
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Bottrop
  - Research Site, Bremen
  - Research Site, Celle
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Erfurt
  - Research Site, Esslingen am Neckar
  - Research Site, Frankfurt (Oder)
  - Research Site, Freiburg i.Br.
  - Research Site, Freital
  - Research Site, Fürth
  - Research Site, Gauting
  - Research Site, Georgsmarienhütte
  - Research Site, Goslar
  - Research Site, Göttingen
  - Research Site, Greifenstein
  - Research Site, Güstrow
  - Research Site, Gütersloh
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidenheim
  - Research Site, Herne
  - Research Site, Hildesheim
  - Research Site, Hof
  - Research Site, Kaiserslautern
  - Research Site, Karlsruhe
  - Research Site, Kempten
  - Research Site, Koblenz
  - Research Site, Krefeld
  - Research Site, Landshut
  - Research Site, Lebach
  - Research Site, Leipzig
  - Research Site, Löwenstein
  - Research Site, Ludwigsburg
  - Research Site, Mainz
  - Research Site, Mönchengladbach
  - Research Site, Muehlheim A.d. Ruhr
  - Research Site, München
  - Research Site, Münnerstadt
  - Research Site, Naunhof
  - Research Site, Neustadt a.R.
  - Research Site, Nuremberg
  - Research Site, Offenburg
  - Research Site, Oldenburg
  - Research Site, Osnabrück
  - Research Site, Pirna
  - Research Site, Porta Westfalica
  - Research Site, Ratingen
  - Research Site, Ravensburg
  - Research Site, Rosenheim
  - Research Site, Rostock
  - Research Site, Schorndorf
  - Research Site, Stolberg
  - Research Site, Stuttgart
  - Research Site, Twistringen
  - Research Site, Völklingen
  - Research Site, Wangen
  - Research Site, Westerstede
  - Research Site, Wiesbaden
  - Research Site, Witten
  - Research Site, Würselen
  - Research Site, Würzburg
  - Research Site, Zittau

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160R00005&attachmentIdentifier=8806c923-cd90-4b13-80a5-000a53f41b0d&fileName=D5160R00005_PANORAMA_Redacted.pdf&versionIdentifier=